CLINICAL TRIAL: NCT02372630
Title: The Effect of TRADJENTA ® (LINAGLIPTIN) on Inflammation, Oxidative Stress and Insulin Resistance in Obese Type 2 Diabetes Subjects
Brief Title: The Effect of LINAGLIPTIN on Inflammation, Oxidative Stress and Insulin Resistance in Obese Type 2 Diabetes Subjects
Acronym: 1971
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University at Buffalo (Other)
Collaborators: Kaleida Health (Other)
Responsible Party: Principal Investigator, Paresh Dandona, Principal Investigator, University at Buffalo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 514091
Record Dates: First submitted 2015-02-20; First posted 2015-02-26 (Estimated); Results first posted 2023-02-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-01

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Linagliptin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Patients will be treated for 12 weeks with placebo once daily
  Interventions: Drug: Placebo
- Linagliptin 5mg per day (Active Comparator): Patients will be treated for 12 weeks with Linagliptin 5mg once daily.
  Interventions: Drug: Linagliptin

INTERVENTIONS:
Drug: Linagliptin — 5 mg daily oral tablets of linagliptin
  Other Names: TRADJENTA
  Arms: Linagliptin 5mg per day
Drug: Placebo — matching placebo giving orally daily
  Arms: Placebo

SUMMARY:
This is a single center, prospective randomized double blind, parallel and placebo controlled study to evaluate oxidative stress and inflammation before and after treatment with linagliptin for 12 weeks. We will also, testing whether Linagliptin is an insulin sensitizer.

DETAILED DESCRIPTION:
This is a single center, prospective randomized double blind, parallel and placebo-controlled study to evaluate oxidative stress and inflammation before and after treatment with linagliptin for 12 weeks. The study enrolls type 2 patients with diabetes.

ELIGIBILITY:
Inclusion Criteria:

Age 20-80 years inclusive. Type 2 diabetes BMI ≥30 kg/m2 Subjects on statins, ACE inhibitors, thiazolidinediones and antioxidants will be allowed as long as they are on stable doses of these compounds and the dosage in not changed during the course of study.

HbA1c ≤ 8.0%

Exclusion Criteria:

- Use of GLP-1 agonists or DPP-IV therapy in the last 3 months. History of Pancreatitis. Risk for pancreatitis, i.e., history of gallstones, alcohol abuse, and hypertriglyceridemia.

Subjects who are taking antiplatelet or anticoagulant medications will be excluded from the fat biopsy portion of the study.

Coronary event or procedure (myocardial infarction, unstable angina, coronary artery bypass, surgery or coronary angioplasty) in the previous four weeks Hepatic disease (liver function tests more than 3 times the upper limit of normal) Renal impairment (serum eGFR <30 ml/min) Any other life-threatening, non-cardiac disease Uncontrolled hypertension (BP > 160/100 mm of Hg) Congestive Heart Failure class III or IV. Use of an investigational agent or therapeutic regimen within 30 days of study Participation in any other concurrent clinical trial

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-05-23 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-05-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- ECMC Ambulatory Center, 3rd Floor, Buffalo, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Patients will be treated for 12 weeks with placebo once daily
  Placebo
- Linagliptin 5mg Per Day: Patients will be treated for 12 weeks with Linagliptin 5mg once daily.
  Linagliptin
Period: Overall Study
Arm/Group | Placebo | Linagliptin 5mg Per Day
Started | 20 | 20
Completed | 17 | 17
Not Completed | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Linagliptin 5mg Per Day | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.9 (10) | 60.8 (8.3) | 59.85 (9.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 11 | 19
  Male | 12 | 9 | 21
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40
BMI [Mean (Standard Deviation); unit: kg/m²] | 37.6 (6.9) | 34.6 (4.8) | 36.1 (5.85)

OUTCOME MEASURES:

1. Primary Outcome: JNK-1 Protein in MNC
Description: JNK-1 protein in MNC before and after linagliptin use as compared to placebo.
Time Frame: Week 0, Week 2, Week 4, Week 12
Measure: Mean (Standard Error); unit: Arbitrary Units
Arm/Group | Placebo | Linagliptin 5mg Per Day
Number analyzed (Participants) | 17 | 17
Arbitrary Units
  Week 0 | 0.943 (0.148) | 0.801 (0.129)
  Week 2 | 1.106 (0.214) | 0.789 (0.101)
  Week 4 | 1.933 (0.204) | 0.702 (0.102)
  Week 12 | 0.939 (0.123) | 0.550 (0.074)

2. Secondary Outcome: IL-1β mRNA Levels
Description: Comparing IL-1B between Linagliptin group and placebo group based on the PCR test, between week 0 and week 12.
Time Frame: Week 0, Week 2, Week 4, Week 12
Measure: Mean (Standard Error); unit: Arbitrary Units
Arm/Group | Placebo | Linagliptin 5mg Per Day
Number analyzed (Participants) | 17 | 17
Arbitrary Units
  Week 0 | 0.768 (0.161) | 1.276 (0.267)
  Week 2 | 0.885 (0.210) | 1.166 (0.240)
  Week 4 | 0.736 (0.144) | 1.063 (0.227)
  Week 12 | 0.811 (0.196) | 0.870 (0.252)

3. Secondary Outcome: Oxidative Stress (as ROS Generation Level)
Description: oxidative stress (ROS generation level) following linagliptin. ROS generation measurement by chemiluminescence of PMN cells
Time Frame: Week 0, Week 2, Week 4, Week 12
Measure: Mean (Standard Error); unit: mV
Arm/Group | Placebo | Linagliptin 5mg Per Day
Number analyzed (Participants) | 17 | 17
mV
  Week 0 | 102 (13) | 91 (8)
  Week 2 | 95 (13) | 85 (11)
  Week 4 | 94 (11) | 81 (8)
  Week 12 | 97 (10) | 76 (8)

4. Secondary Outcome: Insulin Sensitivity by Hyperinsulinemic-euglycemic Clamp
Description: Insulin sensitivity is measured with HE clamp. Glucose Infusion Rate was titrated to maintain blood glucose concentration at the fasting glucose level. Plasma samples for glucose was obtained at 10-minute intervals starting 30 minutes before the clamp, to quantitate rates of whole-body glucose disposal. Difference from baseline at 12 weeks is calculated and compared to placebo arm
Time Frame: At baseline and week 12
Measure: Mean (Standard Error); unit: mL/hr
Arm/Group | Placebo | Linagliptin 5mg Per Day
Number analyzed (Participants) | 17 | 17
mL/hr
  Baseline | 123 (21) | 137 (22)
  At 12 Weeks | 119 (20) | 141 (31)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Placebo | Linagliptin 5mg Per Day
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 0/17 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-05-22): https://cdn.clinicaltrials.gov/large-docs/30/NCT02372630/Prot_SAP_000.pdf